CLINICAL TRIAL: NCT03480464
Title: App-technology to Increase Physical Activity After Bariatric Surgery: A Randomized Controlled Trial
Brief Title: App-technology to Improve the Level of Physical Activity After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Vrinnevi Hospital (Other); Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Ylva Trolle Lagerros, MD, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Dnr: 2016/1259-31/4
Record Dates: First submitted 2017-09-06; First posted 2018-03-29 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Obesity; Bariatric Surgery; Exercise; Quality of Life; Eating Behavior; Body Fat Distribution; Body Weight Changes
MeSH Terms: conditions — Obesity; Motor Activity; Feeding Behavior; Body Weight Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App-technology group (Experimental): App-technology to increase physical activity Participants in the intervention group (App-technology) will use a newly developed smartphone application ("app") in which the participants are able to register their daily physical activity in bouts of 10 min and their intake if supplementary vitamins. They will also be able to set personal goals every week for the level (minutes) of physical activity and get feedback every week in whether they fulfilled the goal or not. They will also get feedback on the intake of supplementary vitamin intake.
  Interventions: Behavioral: App-technology to increase physical activity
- Control group (No Intervention): The control group will receive standard information about the benefit of physical activity after surgery.

INTERVENTIONS:
Behavioral: App-technology to increase physical activity — The application will send daily reminders to register and notices with information about the health benefit of physical activity, medication, supplementary vitamins and diet after surgery
  Other Names: PromMera
  Arms: App-technology group

SUMMARY:
The aim of this study is to investigate the effect of using new app-based technology to increase the level of physical activity, compared to conventional postoperative information given to patients undergoing bariatric surgery. The hypothesis is that the intervention, i.e. using the new technology, will have a greater positive effect on levels of physical activity and outcomes of weight loss than conventional postoperative information.

ELIGIBILITY:
Inclusion Criteria:

* Accepted to bariatric surgery due to national guidelines, BMI>35 kg/m2
* 18 years of age or older
* Informed consent
* Ability to read and understand Swedish
* Own and use a smartphone

Exclusion Criteria:

* Disability preventing daily walking

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Physical activity level | Before surgery and 18 weeks, 6 months, 1 year, and 2 years after surgery.
  counts/min from accelerometers

SECONDARY OUTCOMES:
Body Mass Index | Before surgery, 6 weeks(intervention start) and 18 weeks, 6 months and 1 year after surgery.
  BMI, kg/m2
Body weight | Before surgery, 6 weeks(intervention start) and 18 weeks, 6 months, 1 year, and 2 years after surgery.
  kg
Percent Body Fat | Before surgery, 6 weeks(intervention start) and 18 weeks, 6 months and 1 year after surgery.
  Percent body fat of total body weight
Fat free mass | Before surgery, 6 weeks(intervention start) and 18 weeks, 6 months and 1 year after surgery.
  kg
Muscle mass | Before surgery, 6 weeks(intervention start) and 18 weeks, 6 months and 1 year after surgery.
  kg
Total body water | Before surgery, 6 weeks(intervention start) and 18 weeks, 6 months and 1 year after surgery.
  kg
Hand grip | Before surgery, 6 weeks(intervention start) and 18 weeks, 6 months and 1 year after surgery.
  kg
Self registered physical activity in the app | 12 weeks, 6 to 18 weeks after surgery
  minutes/day and minutes/week

OTHER OUTCOMES:
Change in eating behavior using the TFEQ-R21 questionnaire | Before surgery and 18 weeks, 6 months, 1 year, and 2 years after surgery.
  Eating behavior
Change in Quality of life using the SF35 questionnaire | Before surgery and 18 weeks, 6 months, 1 year, and 2 years after surgery.
  Health related Quality of LIfe
Change in co morbidity, before surgery compared to 1 year and 2 years after surgery. | Before and 1 year and 2 years after surgery
  Number of co morbidities
Change in supplementary vitamin intake adherence according to to the MARS-5 scale | 18 weeks (after surgery) and 1 year after surgery
  Total MARS-5 score, 5-items, 5-point Likert-scale
Change in supplementary vitamin intake adherence using registry data | 18 weeks (after surgery) and 1 year after surgery
  Medication possession ratio, i.e. proportion of fulfilled prescriptions
Change in beliefs and attitude to medication according to the Brief Medication Questionnaire | 18 weeks (after surgery) and 1 year after surgery
  Total BMQ-score, 10 items, 5-point Likert-scale
Change in sleeping habits | Before surgery and 18 weeks, 6 months, 1 year, and 2 years after surgery.
  Assessed using a modified 13-item Karolinska Sleep questionnaire (KSQ)
Change in dietary intake and eating habits | Before surgery and 6 months, 1 year, and 2 years after surgery.
  Macro- and micro-nutrient intake assessed using a 94 item food frequency questionnaire (FFQ)
Change in symptoms related to urinary incontinence or prolapse | Before surgery and 18 weeks, 6 months, 1 year, and 2 years after surgery.
  Assessed using six questions based on the International Consultation on Incontinence Questionnaire
Hemoglobin (Hb) | Before surgery and 1 year after surgery
  g/L
Iron status | Before surgery and 1 year after surgery
  µmol/L
s-folate | Before surgery and 1 year after surgery
  nmol/L
p-calcium | Before surgery and 1 year after surgery
  mmol/L
s-albumin | Before surgery and 1 year after surgery
  g/L
s-cobolamin | Before surgery and 1 year after surgery
  pmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Ylva Trolle Lagerros, Md,PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Vrinnevi Hospital, Norrköping, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bonn SE, Hult M, Spetz K, Eke H, Andersson E, Wiren M, Lof M, Trolle Lagerros Y. Effect of a Smartphone Application on Physical Activity and Weight Loss After Bariatric Surgery-Results from a Randomized Controlled Trial. Obes Surg. 2023 Sep;33(9):2841-2850. doi: 10.1007/s11695-023-06753-6. Epub 2023 Jul 27. PMID 37500930
- [Derived] Spetz K, Hult M, Olbers T, Bonn S, Svedjeholm S, Lagerros YT, Andersson E. A smartphone application to improve adherence to vitamin and mineral supplementation after bariatric surgery. Obesity (Silver Spring). 2022 Oct;30(10):1973-1982. doi: 10.1002/oby.23536. Epub 2022 Sep 1. PMID 36050801
- [Derived] Bonn SE, Hult M, Spetz K, Lof M, Andersson E, Wiren M, Trolle Lagerros Y. App Technology to Support Physical Activity and Intake of Vitamins and Minerals After Bariatric Surgery (the PromMera Study): Protocol of a Randomized Controlled Clinical Trial. JMIR Res Protoc. 2020 Aug 14;9(8):e19624. doi: 10.2196/19624. PMID 32795990